CLINICAL TRIAL: NCT04320355
Title: Exploring the Effects of Soft Tissue Manual Therapy on the Viscoelastic Properties, Pressure Sensitivity and Touch Sensitivity of the Caesarean Section Scar
Brief Title: Exploring the Effects of Soft Tissue Manual Therapy on Caesarean Section Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Interdisciplinary Network Complementary & Alternative Medicine Research (Other); Société Européenne de Recherche en Ostéopathie Pédiatrique et Périnatale (SEROPP) (Unknown)
Responsible Party: Principal Investigator, Isabelle Gilbert, Principal investigator, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-3351
Record Dates: First submitted 2020-03-14; First posted 2020-03-25 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Cesarean Section Complications
Keywords: Caesarean; Manual therapy; Thresholds; Viscoelastic properties; scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: An exploratory descriptive design with before and after measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soft tissue manual therapy (Experimental): The researcher student will place the gloves with the force sensor on the thumb of her right and left hand. She will evaluate the Caesarean section scar and identify the most rigid scar areas when compression is applied. On these identified areas, the researcher student will apply the manual therapy procedure described in the independent variable (compression + shear) section. This procedure will be applied to all identified rigid areas of the Caesarean section scar.This procedure will last 10 minutes (approximately 2 minutes per rigid area). After this time, the researcher-student will remove the force sensor and leave the room.
  Interventions: Other: Soft tissue manual therapy

INTERVENTIONS:
Other: Soft tissue manual therapy — The intervention is a type of massage.

SUMMARY:
Introduction: Caesarean section is one of the most common inpatient surgical procedures. Complications of obstetric wounds are estimated to account for 2.8-26.6% of cases. Between 11 and 15% of women would develop pain and discomfort following a Caesarean section. Manual therapies may be an interesting non-pharmacological approach to treating the signs and symptoms of scarring complications following a Caesarean section. However, the current literature with an in vivo perspective remains modest results for the effects of tissue physiology and their effects on pain.

Method: Using an exploratory "proof of concept" type descriptive design with before and after measurements, the immediate and 7-day effects following the application of soft tissue manual therapy on the Caesarean section scar will be evaluated. The objectives are to describe and explore differences from the effects of soft tissue manual therapy on the viscoelastic properties, pressure sensitivity and touch sensitivity of the Caesarean section scar. Thirty-eight women aged between 18 and 40 years with a Caesarean section scar who attend first-line or specialized obstetrics and perinatal clinics will be recruited.

Anticipated results This project will document the viscoelastic characteristics, pressure sensitivity and touch sensitivity of the C-section scar and surrounding unhealed tissue to improve our understanding of the plausibility of the effects of manual therapy, an approach used to treat the signs and symptoms associated with C-section scarring.

DETAILED DESCRIPTION:
Methods of manual treatment of scars have demonstrated some effectiveness, although the effects and physiology by which mechanical forces of the therapist's hand provide benefits are poorly understood. This research will improve understanding of certain tissue characteristics and physiology elicited during treatment, and provide better conceptual explanations of the effects of manual therapies.

This study consists of 2 steps. The first step consists of the reliability of the Myoton Pro. The second step consists to describe and explore the effects of the soft tissue manual therapy on viscoelastic properties, touch sensibility and pressure sensibility on the Caesarean scar and the unscarred skin.

Objective(s)

The main objective of this project is to evaluate the effects of the application of mechanical force by the therapist's hand on the Caesarean section scar. The specific objectives are to document the following, prior to and following the application of mechanical force by the therapist's hand:

1. Determine the reliability and discrimination of the Myoton Pro.
2. The viscoelastic properties of the Caesarean section scar and surrounding healthy tissues;
3. The sensitivity of the Caesarean section scar to pressure compared with surrounding healthy tissues;
4. The touch sensitivity of the Caesarean section scar compared with surrounding healthy tissue; and
5. Differences in viscoelastic properties, pressure sensitivity and touch sensitivity before and after the independent variable.

Recruitment Recruitment will be recruited women attending primary care and specialized obstetrics and perinatal clinics in the Vaudreuil-Soulanges region, Candiac on the south shore of Montreal, Repentigny located in the Lanaudière region and community organizations with a perinatal orientation located in the Montreal region. Posters will be put up and announcements will be made on the research centre's Facebook page as well as the page dedicated to the project. Interested will be able to communicate directly with the student researcher via digital platform. A brief description of the implications will be sent using digital platform. They will then be asked if they are still interested in participating and if they agree to be contacted by the student researcher in order to verify the eligibility criteria. The student-researcher will request contact information such as email address and a valid telephone number in order to make contact. During this telephone contact, the student-researcher will explain the elements of the study, reiterate the free nature of their participation and verify the eligibility criteria. The student-researcher will then suggest an appointment.

Data collection Phase 1: Reliability of the Myoton Pro The experimental procedure will take place at the Longueuil Campus of the Université de Sherbrooke located in Longueuil. Three evaluators will perform the measurements. The investigator will call them Evaluator 1 (E1), Evaluator 2 (E2) and Evaluator 3 (E3). E1 will invite participants to lie supine on a treatment table. E1 will place a pillow under the participants' knees to reduce the lower extremity strain. They will be asked to undress their abdomen to make the scar visible. The E1 will locate a point in the centre of the scar and a healthy control point about 2 cm above the scar and identify them with an indelible black pencil. The E1 will take four measurements of each point alternately using the MyotonPro. E2 will then take four measurements at the same points using the MyotonPro using the same procedure. Finally, this procedure will be repeated by E3.

Phase 2:

The experimental procedure will take place at the AXiO sports medicine clinic in Vaudreuil-Dorion, the FDL massage therapy and osteopathy clinic located in Candiac, the Parent-aise osteopathy clinic located in Repentigny and the ENOSI osteopathy centre located in Montreal. Measurements of the dependent variables with the MyotonPro, Von Frey's algometer and microfilaments will be taken by a research assistant. She will be trained beforehand on the following elements: 1) the use of Von Frey's microfilaments, 2) the use of the algometer, 3) the use of the Myoton Pro, 4) their application on the tissue and scar points previously identified by the student researcher, 5) computer data entry. The POSAS questionnaire will be administered by the student researcher, who will explain it to the participants.

Upon their arrival, participants will be greeted by the student researcher. The student researcher will give them the consent form, reiterate the free and informed nature of the questionnaire and make sure they understand it. She will ensure that the form is signed. She will then give them the POSAS questionnaire to which will be annexed to the socio-demographic and clinical data questionnaire.

The student-researcher will invite the participants into a room and they will then lie supine on a treatment table. She will then invite the participants to undress the lower abdominal area. The student-researcher will make sure that the Caesarean section scar and the area around it are clearly visible. She will place a pillow under the participants' knees for maximum reduction of any tension surrounding the scar, which will lengthen the lower limbs.

The student-researcher will identify five points on the Caesarean scar, five points on the upper scar border, five points on the lower scar border and five additional points about 2 cm above the scar in the healthy surrounding tissue and mark them with a nontoxic pencil. She will then leave the room.

Using Von Frey's microfilaments, the research assistant will make an initial assessment of the sensitivity to touch of the five points of the Caesarean scar and the healthy tissue. Using the Myoton Pro, the research assistant will make an initial measurement of the viscoelastic properties of the healthy, scarred tissue points and the upper and lower scar edges (for a total of 20 points). Then, the research assistant will use the algometer placed perpendicularly to each identified point and will make a first measurement of pressure sensitivity on the surrounding tissue surfaces and on the Caesarean section scar (T0). In order to ensure reproducibility, 3 measurements per point will be taken before the manual technique is applied. The measurements will be recorded in the participant's file, without the knowledge of the student researcher.

The student-researcher will enter the room. She will place the glove with the force sensor on the thumb of her right hand. She will evaluate the Caesarean section scar and identify the most rigid scar areas when compression is applied. In these identified areas, the student-researcher will apply the manual therapy procedure described in the independent variable (compression + shear) section. This procedure will be applied to all identified rigid areas of the Caesarean section scar.

This procedure will take 20 minutes (approximately 2 minutes per rigid area). After this time, the student-researcher will remove the force sensor and leave the room. The research assistant will perform the evaluation of Von Frey's microfilaments, measurements of viscoelastic properties using the Myoton pro and pressure sensitivity using the algometer at the same tissue and scar points (T1). This same procedure will be performed again seven days later, before (T2) and after the procedure (T3). Following the last measurement time, a complete treatment of the scar area and surrounding tissues will be offered to the participants. Note that an anonymous code will be assigned to each participant and their information. The research assistant will collect the data using an Excel file. The data from the MyotonPro will be collected and automatically saved in a computer folder and later merged into the Excel file.

Sampling The sample of the accessible population will be drawn from a non-probabilistic convenience sample.

Sample size

Phase 1:

The sample size was determined by assuming a predetermined intra-participant standard deviation (Bland and Altman, 1996). Using Bland's formula for repeatability studies, the following parameters were considered: 1) an intra-participant standard deviation of 10%; 2) four measurements at a point on the scar and four measurements at a healthy control point two centimetres above the scar per participant and per evaluator; and 3) three evaluators. Using these parameters, the sample size required to estimate the magnitude of the 95% confidence interval of the precision estimates is 18 participants.

Phase 2:

The exploratory component of this project will provide data with respect to viscoelastic properties, and sensitivity to pressure and touch. Since to our knowledge, no study could inform the sample size calculation, the investigator assume a medium effect size with a power of 80% and a type I error of 5%. Given these assumptions, the sample size requires 32 participants. Anticipating a 10% drop-out rate, the resulting total sample size is 38 participants.

Analysis plan

Phase 1:

In order for the intraclass correlation coefficient (ICC) to be established accurately, the prerequisites of the analysis of variance (ANOVA) must be met. The normality of the observations will be checked using the Kolmogorov-Smirnov test. Using a two-factor ANOVA, the intra-participant standard deviation, repeatability coefficient and ICC will be calculated to establish intra- and inter-rater reliability.

Phase 2:

Descriptive analyses will be conducted based on socio-demographic data and the characteristics of the participants. The continuous variables, if normally distributed, will be summarized using means and standard deviation. The continuous variables, if not normally distributed, will be summarized using medians and intervals. Ordinal and discrete variables will be summarized using percentages.

With respect to the Caesarean section scar, the viscoelastic properties and sensitivity to pre- and post-pressure will be compared using a multi-level longitudinal regression model, if data is normally distributed. Otherwise, nonparametric tests will be performed. The pre- and post-intervention touch sensitivity of the Caesarean section scar will be compared using the Friedman test. A student's paired test will be used to compare POSAS, viscoelastic properties and pressure sensitivity of healthy tissues means. The Wilcoxon rank test will be used for the touch sensitivity of healthy tissues. Finally, the comparison between the Caesarean scar and healthy tissues will be made with the student's test in the case of a normal distribution of data. Otherwise, a nonparametric test will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Woman with a caesarean section scar of 6 months or more but less than two years old
2. with one or more caesarean sections
3. between the ages of 18 and 40
4. with a Pfannenstiel or transverse caesarean section.

Exclusion Criteria:

1. one of the following pathologies: diabetes or under treatment for cancer
2. on anti-inflammatory medication at the time of data collection or they have taken this type of medication in the month prior to data collection
3. applied a product or cream to their scar on the day of data collection
4. contraindications to their skin inductions
5. had a treatment (e.g., a treatment to prevent the development of cancer)
6. undergoing treatment (e.g. laser, massage or other local intervention) for their scar in the three months prior to the data collection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Viscoelastic properties: Stiffness | The change in stiffness is evaluated before and after the intervention. To evaluate this change, two visits each 7 days are required. Stiffness will be assessed at the beginning of each visit and following the intervention.
  The MyotonPro allows the evaluation of five parameters. Stiffness (N/m) is manifested by the resistance to deformation induced by the applied force of the external mechanical arm.The MyotonPro is a portable device that induces a low-force external impulse from a small mechanical external arm. The pulse induces soft tissue oscillations. These are transformed under the force of an acceleration signal and allow the calculation of mechanical and viscoelastic tissue properties.
The viscoelastic properties: Elasticity | The change in Elasticity is evaluated before and after the intervention. To evaluate this change, two visits each 7 days are required. Elasticity will be assessed at the beginning of each visit and following the intervention.
  The MyotonPro allows the evaluation of five parameters. The MyotonPro is a portable device that induces a low-force external impulse from a small mechanical external arm. The pulse induces soft tissue oscillations. These are transformed under the force of an acceleration signal and allow the calculation of mechanical and viscoelastic tissue properties. The ability of the tissue to return to its initial shape characterises elasticity (D). This can be identified by the logarithmic decrement, i.e. the logarithmic measurement of the dissipation of mechanical energy induced by the external arm of the MyotonPro.
The viscoelasticity properties: Tone | The change in tone is evaluated before and after the intervention. To evaluate this change, two visits each 7 days are required. Tone will be assessed at the beginning of each visit and following the intervention.
  The MyotonPro is a portable device that induces a low-force external impulse from a small mechanical external arm. The pulse induces soft tissue oscillations. These are transformed under the force of an acceleration signal and allow the calculation of mechanical and viscoelastic tissue properties. The MyotonPro allows the evaluation of five parameters. The oscillation frequency (Hz) characterizes the resting tone, i.e. the intrinsic cell tension.

SECONDARY OUTCOMES:
Pressure sensitivity | The change in pressure is evaluated before and after the intervention. To evaluate this change, two visits each 7 days are required. Pressure will be assessed at the beginning of each visit and following the intervention.
  Pressure sensitivity rate
Touch sensitivity | The change in touch sensitivity is evaluated before and after the intervention. To evaluate this change, two visits each 7 days are required. Touch sensitivity will be assessed at the beginning of each visit and following the intervention.
  Touch sensitivity rate
Appearance of the caesarean section | The change in appearance is evaluated before the intervention. To evaluate this change, two visits each 7 days are required. Appearance will be assessed at the beginning of each visit.
  Subjective assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nathaly NG Gaudreault, Ph. D, Pt, Study Director — Université de Sherbrooke
Locations (4):
- Canada (4):
  - Clinique d'ostéopathie et de massothérapeie FDL, Candiac, Quebec
  - ENOSI centre d'ostéopathie, Montreal, Quebec
  - Clinide d'ostéopathie Parent-Aise, Repentigny, Quebec
  - AXiO Medecine Clinic, Vaudreuil-Dorion, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adcock D, Paulsen S, Davis S, Nanney L, Shack RB. Analysis of the cutaneous and systemic effects of Endermologie in the porcine model. Aesthet Surg J. 1998 Nov-Dec;18(6):414-20. doi: 10.1016/s1090-820x(98)70069-x. PMID 19328171
- [Background] Al-Benna S, Al-Ajam Y, Tzakas E. Superficial fascial system repair: an abdominoplasty technique to reduce local complications after caesarean delivery. Arch Gynecol Obstet. 2009 May;279(5):673-5. doi: 10.1007/s00404-008-0802-5. Epub 2008 Sep 23. PMID 18810475
- [Background] Bartholomew, S., Deb-Rinker, P., Dzakpasu, S., Système canadien de surveillance périnatale, et Public Health Agency of Canada. (2015). Indicateurs de la santé périnatale au Canada 2013 : Un rapport du Système canadien de surveillance périnatale.
- [Background] Arora PD, Narani N, McCulloch CA. The compliance of collagen gels regulates transforming growth factor-beta induction of alpha-smooth muscle actin in fibroblasts. Am J Pathol. 1999 Mar;154(3):871-82. doi: 10.1016/s0002-9440(10)65334-5. PMID 10079265
- [Background] Beyaz SG, Ozocak H, Ergonenc T, Palabiyik O, Tuna AT, Kaya B, Erkorkmaz U, Akdemir N. Chronic postsurgical pain and neuropathic symptoms after abdominal hysterectomy: A silent epidemic. Medicine (Baltimore). 2016 Aug;95(33):e4484. doi: 10.1097/MD.0000000000004484. PMID 27537570
- [Background] Beyene RT, Kavalukas SL, Barbul A. Intra-abdominal adhesions: Anatomy, physiology, pathophysiology, and treatment. Curr Probl Surg. 2015 Jul;52(7):271-319. doi: 10.1067/j.cpsurg.2015.05.001. Epub 2015 Jun 9. No abstract available. PMID 26258583
- [Background] Bizzini M, Mannion AF. Reliability of a new, hand-held device for assessing skeletal muscle stiffness. Clin Biomech (Bristol). 2003 Jun;18(5):459-61. doi: 10.1016/s0268-0033(03)00042-1. PMID 12763442
- [Background] Bland JM, Altman DG. Measurement error. BMJ. 1996 Jun 29;312(7047):1654. doi: 10.1136/bmj.312.7047.1654. No abstract available. PMID 8664723
- [Background] Bouffard NA, Cutroneo KR, Badger GJ, White SL, Buttolph TR, Ehrlich HP, Stevens-Tuttle D, Langevin HM. Tissue stretch decreases soluble TGF-beta1 and type-1 procollagen in mouse subcutaneous connective tissue: evidence from ex vivo and in vivo models. J Cell Physiol. 2008 Feb;214(2):389-95. doi: 10.1002/jcp.21209. PMID 17654495
- [Background] Brandsborg B, Dueholm M, Kehlet H, Jensen TS, Nikolajsen L. Mechanosensitivity before and after hysterectomy: a prospective study on the prediction of acute and chronic postoperative pain. Br J Anaesth. 2011 Dec;107(6):940-7. doi: 10.1093/bja/aer264. Epub 2011 Sep 2. PMID 21890662
- [Background] Buhimschi CS, Buhimschi IA, Yu C, Wang H, Sharer DJ, Diamond MP, Petkova AP, Garfield RE, Saade GR, Weiner CP. The effect of dystocia and previous cesarean uterine scar on the tensile properties of the lower uterine segment. Am J Obstet Gynecol. 2006 Mar;194(3):873-83. doi: 10.1016/j.ajog.2005.09.004. PMID 16522428
- [Background] Bujold E, Gauthier RJ. Neonatal morbidity associated with uterine rupture: what are the risk factors? Am J Obstet Gynecol. 2002 Feb;186(2):311-4. doi: 10.1067/mob.2002.119923. PMID 11854656
- [Background] Chamorro Comesana A, Suarez Vicente MD, Docampo Ferreira T, Perez-La Fuente Varela MD, Porto Quintans MM, Pilat A. Effect of myofascial induction therapy on post-c-section scars, more than one and a half years old. Pilot study. J Bodyw Mov Ther. 2017 Jan;21(1):197-204. doi: 10.1016/j.jbmt.2016.07.003. Epub 2016 Jul 18. PMID 28167179
- [Background] Chen F, Dellalana LE, Gandelman JS, Vain A, Jagasia MH, Tkaczyk ER. Non-invasive measurement of sclerosis in cutaneous cGVHD patients with the handheld device Myoton: a cross-sectional study. Bone Marrow Transplant. 2019 Apr;54(4):616-619. doi: 10.1038/s41409-018-0346-7. Epub 2018 Oct 4. No abstract available. PMID 30287938
- [Background] Cowman MK, Schmidt TA, Raghavan P, Stecco A. Viscoelastic Properties of Hyaluronan in Physiological Conditions. F1000Res. 2015 Aug 25;4:622. doi: 10.12688/f1000research.6885.1. eCollection 2015. PMID 26594344
- [Background] da Silva RC, de Sa CC, Pascual-Vaca AO, de Souza Fontes LH, Herbella Fernandes FA, Dib RA, Blanco CR, Queiroz RA, Navarro-Rodriguez T. Increase of lower esophageal sphincter pressure after osteopathic intervention on the diaphragm in patients with gastroesophageal reflux. Dis Esophagus. 2013 Jul;26(5):451-6. doi: 10.1111/j.1442-2050.2012.01372.x. Epub 2012 Jun 7. PMID 22676647
- [Background] Damon Mok, W. K. L. (2014). Reliability and Asymmetry Profiles of Myotonometric Measurements in Healthy Skeletal Muscles. Journal of Novel Physiotherapies, 05(01).
- [Background] Dellalana LE, Chen F, Vain A, Gandelman JS, Poldemaa M, Chen H, Tkaczyk ER. Reproducibility of the durometer and myoton devices for skin stiffness measurement in healthy subjects. Skin Res Technol. 2019 May;25(3):289-293. doi: 10.1111/srt.12646. Epub 2018 Nov 10. PMID 30414198
- [Background] Deslauriers V, Rouleau DM, Alami G, MacDermid JC. Translation of the Patient Scar Assessment Scale (PSAS) to French with cross-cultural adaptation, reliability evaluation and validation. Can J Surg. 2009 Dec;52(6):E259-63. PMID 20011161
- [Background] Duffy KJ, Flickinger KL, Kristan JT, Repine MJ, Gianforcaro A, Hasley RB, Feroz S, Rupp JM, Al-Baghli J, Pacella ML, Suffoletto BP, Callaway CW. Quantitative sensory testing measures individual pain responses in emergency department patients. J Pain Res. 2017 May 24;10:1241-1253. doi: 10.2147/JPR.S132485. eCollection 2017. PMID 28579822
- [Background] Freedman BR, Bade ND, Riggin CN, Zhang S, Haines PG, Ong KL, Janmey PA. The (dys)functional extracellular matrix. Biochim Biophys Acta. 2015 Nov;1853(11 Pt B):3153-64. doi: 10.1016/j.bbamcr.2015.04.015. Epub 2015 Apr 27. PMID 25930943
- [Background] Geber C, Klein T, Azad S, Birklein F, Gierthmuhlen J, Huge V, Lauchart M, Nitzsche D, Stengel M, Valet M, Baron R, Maier C, Tolle T, Treede RD. Test-retest and interobserver reliability of quantitative sensory testing according to the protocol of the German Research Network on Neuropathic Pain (DFNS): a multi-centre study. Pain. 2011 Mar;152(3):548-556. doi: 10.1016/j.pain.2010.11.013. Epub 2011 Jan 14. PMID 21237569
- [Background] Gracovetsky S. Can fascia's characteristics be influenced by manual therapy? J Bodyw Mov Ther. 2016 Oct;20(4):893-897. doi: 10.1016/j.jbmt.2016.08.011. Epub 2016 Aug 31. PMID 27814871
- [Background] Grinnell F, Zhu M, Carlson MA, Abrams JM. Release of mechanical tension triggers apoptosis of human fibroblasts in a model of regressing granulation tissue. Exp Cell Res. 1999 May 1;248(2):608-19. doi: 10.1006/excr.1999.4440. PMID 10222153
- [Background] Hausse des taux de césariennes et baisse des taux de naissances | ICIS. (2018, avril 19). Consulté 24 mai 2018, à l'adresse https://www.cihi.ca/en/c-section-rates-continue-to-increase-while-birth-rates-decline.
- [Background] Hinz B. The myofibroblast: paradigm for a mechanically active cell. J Biomech. 2010 Jan 5;43(1):146-55. doi: 10.1016/j.jbiomech.2009.09.020. Epub 2009 Oct 3. PMID 19800625
- [Background] Hinz B, Mastrangelo D, Iselin CE, Chaponnier C, Gabbiani G. Mechanical tension controls granulation tissue contractile activity and myofibroblast differentiation. Am J Pathol. 2001 Sep;159(3):1009-20. doi: 10.1016/S0002-9440(10)61776-2. PMID 11549593
- [Background] Humphrey JD, Dufresne ER, Schwartz MA. Mechanotransduction and extracellular matrix homeostasis. Nat Rev Mol Cell Biol. 2014 Dec;15(12):802-12. doi: 10.1038/nrm3896. Epub 2014 Oct 22. PMID 25355505
- [Background] Ingber DE. Mechanobiology and diseases of mechanotransduction. Ann Med. 2003;35(8):564-77. doi: 10.1080/07853890310016333. PMID 14708967
- [Background] Jafari, L., Gaudreault, N., et Langelier, E. (2016). Viscoelasticity, viscoplasticity and mechanobiological response of fibrous tissues : Current concepts. Journal of Bodywork and Movement Therapies, 20(1), 147-148.
- [Background] Kelly-Martin R, Doughty L, Garkavi M, Wasserman JB. Reliability of modified adheremeter and digital pressure algometer in measuring normal abdominal tissue and C-section scars. J Bodyw Mov Ther. 2018 Oct;22(4):972-979. doi: 10.1016/j.jbmt.2018.02.017. Epub 2018 Feb 17. PMID 30368344
- [Background] Kendig CE. What is Proof of Concept Research and how does it Generate Epistemic and Ethical Categories for Future Scientific Practice? Sci Eng Ethics. 2016 Jun;22(3):735-53. doi: 10.1007/s11948-015-9654-0. Epub 2015 May 26. PMID 26009258
- [Background] Khan KM, Scott A. Mechanotherapy: how physical therapists' prescription of exercise promotes tissue repair. Br J Sports Med. 2009 Apr;43(4):247-52. doi: 10.1136/bjsm.2008.054239. Epub 2009 Feb 24. PMID 19244270
- [Background] Kiener, A., Galli, L., Commare, A., Sabbioni, L., Dall'Asta, A., Frusca, T., et Ghi, T. (2017). EP22.04 : Assessment of Caesarean section scar stiffness by ultrasound elastography. Ultrasound in Obstetrics & Gynecology, 50, 359-359.
- [Background] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520
- [Background] Martinez Rodriguez R, Galan del Rio F. Mechanistic basis of manual therapy in myofascial injuries. Sonoelastographic evolution control. J Bodyw Mov Ther. 2013 Apr;17(2):221-34. doi: 10.1016/j.jbmt.2012.08.006. Epub 2012 Sep 20. PMID 23561871
- [Background] Micallef L, Vedrenne N, Billet F, Coulomb B, Darby IA, Desmouliere A. The myofibroblast, multiple origins for major roles in normal and pathological tissue repair. Fibrogenesis Tissue Repair. 2012 Jun 6;5(Suppl 1):S5. doi: 10.1186/1755-1536-5-S1-S5. eCollection 2012. PMID 23259712
- [Background] O'Neill S, O'Neill L. Improving QST Reliability--More Raters, Tests, or Occasions? A Multivariate Generalizability Study. J Pain. 2015 May;16(5):454-62. doi: 10.1016/j.jpain.2015.01.476. Epub 2015 Feb 13. PMID 25683899
- [Background] Pesteil, F., Vignaud, L., Bonté, F., et Desmoulière, A. (2017). Rôles primordiaux des fibroblastes dermiques dans la cicatrisation cutanée. Revue Francophone de Cicatrisation, 1(3), 45-49.
- [Background] Rosinczuk J, Taradaj J, Dymarek R, Sopel M. Mechanoregulation of Wound Healing and Skin Homeostasis. Biomed Res Int. 2016;2016:3943481. doi: 10.1155/2016/3943481. Epub 2016 Jun 20. PMID 27413744
- [Background] Schleip, R. (2003). Fascial plasticity - a new neurobiological explanation Part 2. Journal of Bodywork and Movement Therapies, 7(2), 104-116.
- [Background] Schleip R, Naylor IL, Ursu D, Melzer W, Zorn A, Wilke HJ, Lehmann-Horn F, Klingler W. Passive muscle stiffness may be influenced by active contractility of intramuscular connective tissue. Med Hypotheses. 2006;66(1):66-71. doi: 10.1016/j.mehy.2005.08.025. Epub 2005 Oct 4. PMID 16209907
- [Background] Schneider S, Peipsi A, Stokes M, Knicker A, Abeln V. Feasibility of monitoring muscle health in microgravity environments using Myoton technology. Med Biol Eng Comput. 2015 Jan;53(1):57-66. doi: 10.1007/s11517-014-1211-5. Epub 2014 Oct 21. PMID 25331739
- [Background] Seliger G, Chaoui K, Lautenschlager C, Jenderka KV, Kunze C, Hiller GGR, Tchirikov M. Ultrasound elastography of the lower uterine segment in women with a previous cesarean section: Comparison of in-/ex-vivo elastography versus tensile-stress-strain-rupture analysis. Eur J Obstet Gynecol Reprod Biol. 2018 Jun;225:172-180. doi: 10.1016/j.ejogrb.2018.04.013. Epub 2018 Apr 20. PMID 29729520
- [Background] Silver FH, Ebrahimi A, Snowhill PB. Viscoelastic properties of self-assembled type I collagen fibers: molecular basis of elastic and viscous behaviors. Connect Tissue Res. 2002;43(4):569-80. PMID 12685863
- [Background] Simons GD, Mense S. Understanding and measurement of muscle tone as related to clinical muscle pain. Pain. 1998 Mar;75(1):1-17. doi: 10.1016/S0304-3959(97)00102-4. PMID 9539669
- [Background] Solomonow M, He Zhou B, Baratta RV, Lu Y, Zhu M, Harris M. Biexponential recovery model of lumbar viscoelastic laxity and reflexive muscular activity after prolonged cyclic loading. Clin Biomech (Bristol). 2000 Mar;15(3):167-75. doi: 10.1016/s0268-0033(99)00062-5. PMID 10656978
- [Background] Standley PR. My personal journey that led to the crossroads of interdisciplinary manual medicine research: serendipitous opportunities afforded a basic scientist. J Bodyw Mov Ther. 2013 Jan;17(1):79-82. doi: 10.1016/j.jbmt.2012.08.002. Epub 2012 Sep 7. No abstract available. PMID 23294687
- [Background] Tena B, Escobar B, Arguis MJ, Cantero C, Rios J, Gomar C. Reproducibility of Electronic Von Frey and Von Frey monofilaments testing. Clin J Pain. 2012 May;28(4):318-23. doi: 10.1097/AJP.0b013e31822f0092. PMID 22001670
- [Background] Tulandi T, Agdi M, Zarei A, Miner L, Sikirica V. Adhesion development and morbidity after repeat cesarean delivery. Am J Obstet Gynecol. 2009 Jul;201(1):56.e1-6. doi: 10.1016/j.ajog.2009.04.039. PMID 19576375
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Van De Water L, Varney S, Tomasek JJ. Mechanoregulation of the Myofibroblast in Wound Contraction, Scarring, and Fibrosis: Opportunities for New Therapeutic Intervention. Adv Wound Care (New Rochelle). 2013 May;2(4):122-141. doi: 10.1089/wound.2012.0393. PMID 24527336
- [Background] van der Wal MB, Tuinebreijer WE, Lundgren-Nilsson A, Middelkoop E, van Zuijlen PP. Differential item functioning in the Observer Scale of the POSAS for different scar types. Qual Life Res. 2014 Sep;23(7):2037-45. doi: 10.1007/s11136-014-0637-4. Epub 2014 Feb 9. PMID 24510653
- [Background] Vermillion ST, Lamoutte C, Soper DE, Verdeja A. Wound infection after cesarean: effect of subcutaneous tissue thickness. Obstet Gynecol. 2000 Jun;95(6 Pt 1):923-6. doi: 10.1016/s0029-7844(99)00642-0. PMID 10831993
- [Background] Vranova H, Zeman J, Cech Z, Otahal S. Identification of viscoelastic parameters of skin with a scar in vivo, influence of soft tissue technique on changes of skin parameters. J Bodyw Mov Ther. 2009 Oct;13(4):344-9. doi: 10.1016/j.jbmt.2008.06.004. Epub 2008 Nov 4. PMID 19761958
- [Background] Wasserman, Jennifer B., Abraham, K., Massery, M., Chu, J., Farrow, A., et Marcoux, B. C. (2018). Soft Tissue Mobilization Techniques Are Effective in Treating Chronic Pain Following Cesarean Section : A Multicenter Randomized Clinical Trial. Journal of Women's Health Physical Therapy, 1
- [Background] Wasserman JB, Steele-Thornborrow JL, Yuen JS, Halkiotis M, Riggins EM. Chronic caesarian section scar pain treated with fascial scar release techniques: A case series. J Bodyw Mov Ther. 2016 Oct;20(4):906-913. doi: 10.1016/j.jbmt.2016.02.011. Epub 2016 Mar 10. PMID 27814873
- [Background] Weibel S, Neubert K, Jelting Y, Meissner W, Wockel A, Roewer N, Kranke P. Incidence and severity of chronic pain after caesarean section: A systematic review with meta-analysis. Eur J Anaesthesiol. 2016 Nov;33(11):853-865. doi: 10.1097/EJA.0000000000000535. PMID 27635953
- [Background] Wight TN, Potter-Perigo S. The extracellular matrix: an active or passive player in fibrosis? Am J Physiol Gastrointest Liver Physiol. 2011 Dec;301(6):G950-5. doi: 10.1152/ajpgi.00132.2011. Epub 2011 Apr 21. PMID 21512158
- [Background] Wong VW, Beasley B, Zepeda J, Dauskardt RH, Yock PG, Longaker MT, Gurtner GC. A Mechanomodulatory Device to Minimize Incisional Scar Formation. Adv Wound Care (New Rochelle). 2013 May;2(4):185-194. doi: 10.1089/wound.2012.0396. PMID 24527342
- [Background] Zhang J, Miller CJ, O'Malley V, Bowman EB, Etzkorn JR, Shin TM, Sobanko JF. Patient and Physician Assessment of Surgical Scars: A Systematic Review. JAMA Facial Plast Surg. 2018 Jul 1;20(4):314-323. doi: 10.1001/jamafacial.2017.2314. PMID 29392275
- [Derived] Gilbert I, Gaudreault N, Gaboury I. Exploring the Effects of Standardized Soft Tissue Mobilization on the Viscoelastic Properties, Pressure Pain Thresholds, and Tactile Pressure Thresholds of the Cesarean Section Scar. J Integr Complement Med. 2022 Apr;28(4):355-362. doi: 10.1089/jicm.2021.0178. Epub 2022 Jan 13. PMID 35426735